CLINICAL TRIAL: NCT04409964
Title: the Effect of Opioid-free General Anesthesia on the Recovery Quality After Gynecological Laparoscopy
Brief Title: the Effect of Opioid-free General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Young Eun Moon, associate professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: OFGA
Record Dates: First submitted 2020-05-26; First posted 2020-06-01 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Gynecologic Disease
MeSH Terms: conditions — Genital Diseases, Female | interventions — Dexmedetomidine; Lidocaine; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- opioid-free anesthesia (Experimental): The study group receives the dexmedetomidine and lidocaine infusion with general anesthesia for gynecological laparoscopy.
  Interventions: Drug: Dexmedetomidine Hydrochloride; Drug: Lidocaine Hydrochloride
- opioid anesthesia (Active Comparator): The control group receives the remifentanil infusion with general anesthesia for gynecological laparoscopy.
  Interventions: Drug: Remifentanil Hydrochloride

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride — dexmedetomidine iv bolus followed by the infusion of 0.1-1 ug/kg/hr during general anesthesia
  Other Names: precedex
  Arms: opioid-free anesthesia
Drug: Lidocaine Hydrochloride — lidocaine iv bolus followed by the infusion of 1.5 mg/kg/hr during general anesthesia
  Other Names: lidocaine
  Arms: opioid-free anesthesia
Drug: Remifentanil Hydrochloride — remifentanil iv infusion of 0.5-5 ng/ml (effect site concentration using TCI) during general anesthesia
  Other Names: remifentanil
  Arms: opioid anesthesia

SUMMARY:
This study is performed to investigate the effect of opioid-free general anesthesia on the recovery quality after gynecological laparoscopy.

DETAILED DESCRIPTION:
The quality of recovery after the surgery is assessed using the QoR 40. In addition, the various kinds of cytokine are assessed for the ancillary study.

ELIGIBILITY:
Inclusion Criteria:

* patient scheduled for gynecological laparoscopic surgery

Exclusion Criteria:

1. refusal to participate in this study
2. emergent surgery
3. chronic pain requiring for pain killer
4. psychiatric disease
5. preoperative bradycardia or hypotension
6. allergy or history of the adverse effect to study drug
7. pregnancy or lactation

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — the patients undergoing the gynecological laparoscopic surgery
Enrollment: 78 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
the quality of recovery | at 24 hour after the completion of surgery
  The quality of recovery is assessed using questionnaire. This questionnaire includes 40 items. The score range is from 40 to 200. The higher score means the better quality of recovery after surgery.

SECONDARY OUTCOMES:
cytokine | during surgery
  as ancillary study, to assess the various kinds of cytokines such as epinephrine, norepinephrine, interleukin-10, tumor necrosis factor-alpha.

CONTACTS AND LOCATIONS:
Overall Officials: Youngeun Moon, MD, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul St.Mary's Hospital, Seoul, Seocho-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Song JY, Choi H, Chae M, Ko J, Moon YE. The effect of opioid-free anesthesia on the quality of recovery after gynecological laparoscopy: study protocol for a prospective randomized controlled trial. Trials. 2021 Mar 12;22(1):207. doi: 10.1186/s13063-021-05166-z. PMID 33712080